CLINICAL TRIAL: NCT01841281
Title: Phase II Study of L-arginine in Severe Asthma Patients Grouped by Exhaled Nitric Oxide Level
Brief Title: L-arginine in Severe Asthma Patients Grouped by Exhaled Nitric Oxide Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nicholas Kenyon (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Nicholas Kenyon, Professor, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 271515; R01HL105573 (NIH); UCD105573 (Other: UC Davis)
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Asthma; Inflammation
Keywords: Asthma; Severe Asthma
MeSH Terms: conditions — Asthma; Inflammation | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Exhaled Nitric Oxide (NO) (Active Comparator): Subjects with a baseline exhaled NO level less than or equal to 20 ppb will be enrolled in the Low Exhaled Nitric Oxide arm.
  All subjects will receive L-arginine and placebo in this cross-over design study.
  Interventions: Drug: L-Arginine; Drug: Placebo
- High Exhaled Nitric Oxide (NO) (Active Comparator): Subjects with a baseline exhaled NO level greater than or equal to 25 ppb will be enrolled in the High Exhaled Nitric Oxide arm.
  All subjects will receive L-arginine and placebo in this cross-over design study.
  Interventions: Drug: L-Arginine; Drug: Placebo

INTERVENTIONS:
Drug: L-Arginine — L-arginine tablets containing 1 g of elemental L-arginine (1204 mg of L-arginine HCL) developed by Jarrow Formulas in Los Angeles.
  Other Names: Arginine 1000 (Jarrow Formulas, Los Angeles, CA)
Drug: Placebo — Matching placebo tablets do not contain L-arginine. Placebo tablets were manufactured by Jarrow Formulas and contain cellulose and other excipients.

SUMMARY:
The major impact of this study will be to identify the adult severe asthma cohort that will benefit from supplemental L-arginine therapy. The investigators hypothesize that a subset of adult severe asthma patients will respond to supplemental L-arginine and derive clinical benefit from the addition of this therapy to standard-of-care asthma medications. The investigators hypothesize that the patients that benefit most will have low exhaled nitric oxide concentrations (< 20 ppb) at baseline.

DETAILED DESCRIPTION:
We hypothesize that a subset of adult severe asthma patients will respond to supplemental L-arginine and derive clinical benefit from the addition of this therapy to standard-of-care medications. We hypothesize that these patients will have lower exhaled NO concentrations (<20 ppb) and lower nitric oxide synthase 2 (NOS2)/ arginase I (Arg1) mRNA ratios in their airway epithelial cells than "non-responders." The aim is to test the hypothesis that adult severe asthma subjects with exhaled breath NO concentrations < 20 ppb will have fewer American Thoracic Society (ATS)-defined asthma exacerbations over 3 months when treated with L-arginine compared to subjects with exhaled nitric oxide concentration (FeNO) > 25 ppb. The major impact of this study will be to identify the adult severe asthma cohort that will benefit from supplemental L-arginine therapy to define the underlying mechanisms of arginine benefit in asthma. This follows our initial 20 subject trial of L-arginine in asthma subjects (Kenyon et al., Pharmaceuticals 2011) that was designed to determine how L-arginine was metabolized (by testing serum markers) and whether certain participants had clinical benefit.

To do this, we will recruit a total of 50 ATS-defined severe asthmatic subjects with ongoing asthma exacerbations in past two months and enroll them in a randomized, blinded, placebo-controlled, cross-over designed trial of L-arginine and placebo. We will compare 25 subjects with "low" FeNO < 20 with 25 subjects that have "high" FeNO > 25 ppb.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 yrs of age
* Diagnosis of severe asthma based on American Thoracic Society Workshop definition (Am J Respir Crit Care Med 2000; 162:2341)
* Active asthma medications of high dose inhaled corticosteroids plus long-acting beta agonist
* History of recent asthma exacerbations or Asthma control test score < 20/25

Exclusion Criteria:

* <19 yrs of age
* Forced expiratory volume 1sec <30% predicted
* Pregnant or nursing women
* Current smokers or smoking history > 15 pack years
* Actively taking or known intolerance to L-arginine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-08; Primary Completion 2018-08 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Kenyon, MD,MS, Principal Investigator — Univ. of California, Davis
Locations (1):
- UC Davis CTSC Clinical Research Center, Sacramento, California, United States

REFERENCES:
- [Derived] Liao SY, Showalter MR, Linderholm AL, Franzi L, Kivler C, Li Y, Sa MR, Kons ZA, Fiehn O, Qi L, Zeki AA, Kenyon NJ. l-Arginine supplementation in severe asthma. JCI Insight. 2020 Jul 9;5(13):e137777. doi: 10.1172/jci.insight.137777. PMID 32497023

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 54 subjects consented and enrolled for the trial, but n=50 were randomized as n=4 participants declined to participate.
Pre-assignment Details: Participants were assigned to low or high exhaled nitric oxide groups based on their levels at time of Visit 1.
Groups:
- Low Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo: Subjects with a baseline exhaled NO level less than or equal to 20 ppb
  Receive L-arginine first, then Placebo
  L-Arginine: L-arginine tablets containing 1 g of elemental L-arginine (1204 mg of L-arginine HCL) developed by Jarrow Formulas in Los Angeles.
  Placebo: Matching placebo tablets do not contain L-arginine. Placebo tablets were manufactured by Jarrow Formulas and contain cellulose and other excipients.
- High Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo; High Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine: Subjects with a baseline exhaled NO level greater than or equal to 25 ppb
  Receive L-arginine first, then Placebo
  L-Arginine: L-arginine tablets containing 1 g of elemental L-arginine (1204 mg of L-arginine HCL) developed by Jarrow Formulas in Los Angeles.
  Placebo: Matching placebo tablets do not contain L-arginine. Placebo tablets were manufactured by Jarrow Formulas and contain cellulose and other excipients.
- Low Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine: Subjects with a baseline exhaled NO level less than or equal to 20 ppb
  Receive Placebo first, then L-arginine
  L-Arginine: L-arginine tablets containing 1 g of elemental L-arginine (1204 mg of L-arginine HCL) developed by Jarrow Formulas in Los Angeles.
  Placebo: Matching placebo tablets do not contain L-arginine. Placebo tablets were manufactured by Jarrow Formulas and contain cellulose and other excipients.
Period: First Intervention (12 Weeks)
Arm/Group | Low Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo | High Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo | Low Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine | High Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine
Started | 11 | 12 | 13 | 14
Completed | 11 | 12 | 13 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Washout (6 Weeks)
Arm/Group | Low Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo | High Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo | Low Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine | High Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine
Started | 11 | 12 | 13 | 14
Completed | 9 | 9 | 10 | 13
Not Completed | 2 | 3 | 3 | 1
Period: Second Intervention (12 Weeks)
Arm/Group | Low Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo | High Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo | Low Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine | High Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine
Started | 9 | 9 | 10 | 13
Completed | 9 | 6 | 10 | 13
Not Completed | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Exhaled Nitric Oxide (NO): Subjects with a baseline exhaled NO level less than or equal to 20 ppb will be enrolled in the Low Exhaled Nitric Oxide arm.
  Baseline characteristics at the enrollment
- High Exhaled Nitric Oxide (NO): Subjects with a baseline exhaled NO level greater than or equal to 25 ppb will be enrolled in the High Exhaled Nitric Oxide arm.
  Baseline characteristics at the enrollment
- Total: Total of all reporting groups
Arm/Group | Low Exhaled Nitric Oxide (NO) | High Exhaled Nitric Oxide (NO) | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (11.9) | 52.4 (14.3) | 54.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 7 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 20 | 39
  Non-White | 5 | 6 | 11
Spirometry [Mean (Standard Deviation); unit: Litters]
  FEV1 | 1.8 (0.7) | 2.2 (0.9) | 2 (0.8)
  FVC | 2.6 (0.9) | 2.8 (1.1) | 2.7 (1.0)
Weight [Mean (Standard Deviation); unit: Kg] | 94.8 (20.5) | 85.6 (27.3) | 90.0 (24.5)
Asthma Control Test Score [Mean (Standard Deviation); unit: units on a scale] — The total Asthma Control Test score is reported. It is on a scale of 5 to 25. The higher the score, the better the asthma control. A score of 20 or more suggests good asthma control. A score of less than 20 suggests inadequate asthma control.
  units on a scale | 16.0 (4.6) | 16.1 (5.5) | 16.1 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Acute Exacerbation at 3 Months
Description: The primary endpoint of the study is the number of acute moderate exacerbations at 3 months. A moderate asthma exacerbation is defined as any of the following: 1) A drop in morning peak flow rate (PEFR) >30% from baseline on 2 consecutive days (1 event), 2) Need for initiation of oral steroids or am increased dose of inhaled corticosteroids on any two consecutive days (1 event), 3) Doubling of short-acting β-agonist use (e.g. number of puffs of albuterol) per day for 2 consecutive days (1 event).
Time Frame: 3 month
Population: Several patients dropped after the first intervention
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Low Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo | High Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo | Low Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine | High Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine
Number analyzed (Participants) | 11 | 12 | 13 | 14
Events
  First Intervention | 2.7 (2.0) | 2.2 (2.2) | 1.6 (1.8) | 2.2 (3.0)
  Second Intervention: number analyzed (Participants) | 9 | 6 | 10 | 13
  Second Intervention | 2.1 (1.4) | 2.7 (4.2) | 2.2 (2.2) | 2.2 (2.8)
Statistical Analysis 1: Comparison: Low Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo vs High Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo vs Low Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine vs High Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine; Test type: Other; p = 0.78, testing for interaction term — The p-value is for the interaction term

2. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)/Forced Vital Capacity (FVC)
Description: The secondary endpoint is the change in FEV1/FVC ratio at 3 months. This calcuation is a ratio between the volume of breath exhaled in the first second divided by the total amount of breath exhaled in a vital capacity maneuver. A normal ratio is usually > 70%.
Time Frame: 3 month
Population: Several patients dropped after the first intervention
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo | High Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo | Low Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine | High Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine
Number analyzed (Participants) | 11 | 12 | 13 | 14
ratio
  First Intervention | -0.02 (0.05) | 0.01 (0.06) | 0.03 (0.13) | -0.03 (0.04)
  Second Intervention: number analyzed (Participants) | 9 | 6 | 10 | 13
  Second Intervention | 0.01 (0.04) | 0.13 (0.06) | 0.003 (0.06) | -0.04 (0.10)
Statistical Analysis 1: Comparison: Low Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo vs High Exhaled Nitric Oxide (NO), L-Arginine First, Then Placebo vs Low Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine vs High Exhaled Nitric Oxide (NO), Placebo First, Then L-Arginine; The treatment effect was tested as an interaction term between treatment and FeNO. The null hypothesis is the effect of treatment is stratified by the FeNO status. We used a regression model instead of t-test or Wilcoxon signed-rank test in order to control period and carry-over effect which is common in a cross-over study design; Test type: Other; p = 0.09, testing for interaction term — The p-value is for the interaction term

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the trial,8 months
Groups:
- Low Exhaled Nitric Oxide (NO) Phase 1, Treatment Arm: ow Exhaled Nitric Oxide (NO) Phase 1, L-Arginine arm
- Low Exhaled Nitric Oxide (NO) Phase 1, Placebo Arm: Low Exhaled Nitric Oxide (NO) Phase 1, placebo arm
- Low Exhaled Nitric Oxide (NO) Washout Phase: Low Exhaled Nitric Oxide (NO) Washout Phase
- Low Exhaled Nitric Oxide (NO) Phase 2, Treatment Arm: Low Exhaled Nitric Oxide (NO) Phase 2, L-Arginine arm
- Low Exhaled Nitric Oxide (NO) Phase 2, Placebo Arm: Low Exhaled Nitric Oxide (NO) Phase 2, placebo arm
- High Exhaled Nitric Oxide (NO) Phase 1, Treatment Arm: High Exhaled Nitric Oxide (NO) Phase 1, L-Arginine arm
- High Exhaled Nitric Oxide (NO) Phase 1, Placebo Arm: High Exhaled Nitric Oxide (NO) Phase 1, placebo arm
- High Exhaled Nitric Oxide (NO) Washout Phase: High Exhaled Nitric Oxide (NO) Washout Phase
- High Exhaled Nitric Oxide (NO) Phase 2, Treatment Arm: High Exhaled Nitric Oxide (NO) Phase 2, L-Arginine arm
- High Exhaled Nitric Oxide (NO) Phase 2, Placebo Arm: igh Exhaled Nitric Oxide (NO) Phase 2, Placebo arm
Arm/Group | Low Exhaled Nitric Oxide (NO) Phase 1, Treatment Arm | Low Exhaled Nitric Oxide (NO) Phase 1, Placebo Arm | Low Exhaled Nitric Oxide (NO) Washout Phase | Low Exhaled Nitric Oxide (NO) Phase 2, Treatment Arm | Low Exhaled Nitric Oxide (NO) Phase 2, Placebo Arm | High Exhaled Nitric Oxide (NO) Phase 1, Treatment Arm | High Exhaled Nitric Oxide (NO) Phase 1, Placebo Arm | High Exhaled Nitric Oxide (NO) Washout Phase | High Exhaled Nitric Oxide (NO) Phase 2, Treatment Arm | High Exhaled Nitric Oxide (NO) Phase 2, Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13 | 0/19 | 0/10 | 0/9 | 0/12 | 0/14 | 0/22 | 0/16 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/19 | 0/10 | 0/9 | 2/12 | 1/14 | 1/22 | 0/16 | 0/6
Other Adverse Events (participants affected / at risk) | 0/11 | 1/13 | 0/19 | 1/10 | 0/9 | 1/12 | 0/14 | 0/22 | 0/16 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Exhaled Nitric Oxide (NO) Phase 1, Treatment Arm (N=11) | Low Exhaled Nitric Oxide (NO) Phase 1, Placebo Arm (N=13) | Low Exhaled Nitric Oxide (NO) Washout Phase (N=19) | Low Exhaled Nitric Oxide (NO) Phase 2, Treatment Arm (N=10) | Low Exhaled Nitric Oxide (NO) Phase 2, Placebo Arm (N=9) | High Exhaled Nitric Oxide (NO) Phase 1, Treatment Arm (N=12) | High Exhaled Nitric Oxide (NO) Phase 1, Placebo Arm (N=14) | High Exhaled Nitric Oxide (NO) Washout Phase (N=22) | High Exhaled Nitric Oxide (NO) Phase 2, Treatment Arm (N=16) | High Exhaled Nitric Oxide (NO) Phase 2, Placebo Arm (N=6)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Subject was admitted to the hospital for exacerbation or flare of asthma either on placebo or L-arginine.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Exhaled Nitric Oxide (NO) Phase 1, Treatment Arm (N=11) | Low Exhaled Nitric Oxide (NO) Phase 1, Placebo Arm (N=13) | Low Exhaled Nitric Oxide (NO) Washout Phase (N=19) | Low Exhaled Nitric Oxide (NO) Phase 2, Treatment Arm (N=10) | Low Exhaled Nitric Oxide (NO) Phase 2, Placebo Arm (N=9) | High Exhaled Nitric Oxide (NO) Phase 1, Treatment Arm (N=12) | High Exhaled Nitric Oxide (NO) Phase 1, Placebo Arm (N=14) | High Exhaled Nitric Oxide (NO) Washout Phase (N=22) | High Exhaled Nitric Oxide (NO) Phase 2, Treatment Arm (N=16) | High Exhaled Nitric Oxide (NO) Phase 2, Placebo Arm (N=6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT01841281/Prot_SAP_000.pdf